CLINICAL TRIAL: NCT00918814
Title: A Dose-Ranging and Dose Frequency Study Evaluating the Safety and Efficacy of LIPO-102 for the Reduction of Abdominal Subcutaneous Adipose Tissue
Brief Title: Dose Ranging and Dose Frequency of LIPO-102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIPO-102-CL-03
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Subcutaneous Adipose Tissue Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIPO-102 (Experimental): LIPO-102
  Interventions: Drug: LIPO-102
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-102 — Subcutaneous Injection
  Arms: LIPO-102
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Dose Ranging and Dose Frequency of LIPO-102

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant female
* Good general health
* Sufficient abdominal fat for injections
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to study drugs
* Treatment with an investigational agent within 30 days of first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety: physical examinations, laboratory tests, AE assessment | 4 weeks treatment and 4 weeks follow up

SECONDARY OUTCOMES:
Efficacy: change in subcutaneous abdominal adipose tissue thickness | 4 weeks treatment and 4 weeks follow up

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego, California
  - Baltimore, Maryland